CLINICAL TRIAL: NCT06950762
Title: Aesthetic Performance of Two Injectable Resin Composites in Class V Cavities: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Abdelrhman Elhariry, Principal Investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: class v restoration
Record Dates: First submitted 2025-04-12; First posted 2025-04-30 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Restoration of Carious Class v Anterior Teeth
Keywords: Giomer based injectable composite

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beautifil flow plus x f00 (Active Comparator): Bioactive giomer based injectable resin composite
  Interventions: Procedure: Giomer based injectable composite
- G-aenial universal injectable resin composite (Active Comparator): conventional injectable resin composite
  Interventions: Procedure: Universal injectable resin composite

INTERVENTIONS:
Procedure: Giomer based injectable composite — Giomers utilize surface pre-reacted glass (SPRG) technology, which involves an acid-base reaction between fluorine-containing glass particles and polymer-containing acid when exposed to water. This reaction results in the formation of a glass ionomer phase, which is then dispersed throughout the resin. Furthermore, the S-PRG fillers present in giomer materials enable the continuous release and replenishment of fluoride, offering long-lasting protection against the recurrence of caries
  Arms: Beautifil flow plus x f00
Procedure: Universal injectable resin composite — Conventional injectable resin composite
  Arms: G-aenial universal injectable resin composite

SUMMARY:
Using bioactive injectable resin composite in anterior class v carious lesions can provide better aesthetic outcome and marginal integrity by releasing multiple ions, including fluoride. This offers better marginal integrity due to presence of S-PRG fillers

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-60 years.
2. Co-operative participants approving to participate in the study.
3. Male or female patients.
4. Medically free participants.
5. Moderate or high caries risk participants.

Exclusion Criteria:

1. Systemic disease or severe medical complications.
2. Participants with a history of allergy to any component of restorations will be used in the study.
3. Lack of compliance
4. Evidence of severe bruxism, clenching, or temporomandibular joint disorders or bizarre habits

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Marginal discoloration using FDI criteria | 12 Month

IPD SHARING:
Plan to Share IPD: Yes